CLINICAL TRIAL: NCT06177730
Title: PACER:Pre-hospital ECMO or Conventional Resuscitation for Refractory Cardiac Arrest. An Investigator Initiated, Parallel Group, Assessor-blinded, Registry Embedded, Randomised Controlled Pilot Trial
Brief Title: Pre-hospital ECMO or Conventional Resuscitation for Refractory Cardiac Arrest
Acronym: PACER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Ambulance Victoria (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANZIC-RC/SR001
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: ECMO; OHCA; pre-hospital; Extracorporeal Membrane Oxygenation; Out of Hospital Cardiac Arrest; ECPR; Extracorproreal Membrane Oxygenation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-hospital ECPR Strategy (Active Comparator): All patients will have high performance CPR at the scene throughout the resuscitation. If the patient is randomised to the Pre-hospital ECPR Strategy, this will be continued until the PACER team arrives. If return of spontaneous circulation (ROSC) has not been achieved at this point, ECPR will be implemented. The patient will be transported to The Alfred Hospital to receive ongoing care.
  Interventions: Other: Pre-Hospital ECPR
- Conventional Cardiac Arrest Strategy (No Intervention): All patients will have high performance CPR at the scene throughout the resuscitation. If the patient has been randomised to the Conventional Cardiac Arrest Strategy and ROSC has not occurred after >20 minutes, ongoing resuscitation will occur and the patient may be transported via AV to the nearest emergency cardiac catheterisation capable hospital where conventional resuscitation care will continue and Hospital based ECPR may be implemented if the patient meets local eligibility criteria. This is in line with current practice.

INTERVENTIONS:
Other: Pre-Hospital ECPR — Implementation of pre-Hospital ECPr in OHCA
  Arms: Pre-hospital ECPR Strategy

SUMMARY:
This pilot study aims to determine feasibility of randomising patients to receive pre-hospital Extracorporeal Cardiopulmonary Resuscitation (ECPR) compared to conventional cardiac arrest care for refractory out of hospital cardiac arrest (OHCA).

The success of this study will be measured by the number of patients recruited into the study successfully treated with the treatment they were randomised to receive in the pre-Hospital setting.

DETAILED DESCRIPTION:
Conventional cardiac arrest care, including high performance cardiopulmonary resuscitation, defibrillation and administration of drugs such as adrenaline is the current treatment for out of hospital cardiac arrest. In cases where this treatment does not see spontaneous circulation restored promptly, the patients cardiac arrest is termed refractory. Refractory Cardiac arrest is coupled with an increased risk of hypoxic injury to vital organs and the prospect of survival with good neurological recovery decreases dramatically.

ECPR is an effective way to restore circulation for patients with refractory OHCA. Hospital based ECPR is the most common process by which refractory OHCA patients are treated with ECPR. Patients are transported to an ECPR capable hospital while receiving mechanical CPR. Transporting patients while receiving mechanical CPR is challenging and may lead to less effective CPR (low flow). It may also delay access to urgent hospital based treatments due to the extra time required to load a patient receiving mechanical CPR.

Pre-Hospital ECPR is where the ECMO team rapidly attends the scene and implements ECMO while CPR is on-going at the scene. Benefits of this approach may include reduced low-flow time due to both earlier ECMO initiation as well as allowing the emergency responders focus on delivering high performance CPR rather than loading the patient for transport.

The results of this study will inform a larger study where researchers will compare these two treatments to determine if ECPR leads to higher survival rates and better recovery for patients with refractory OHCA. Observational data for pre-hospital ECPR in the Australian setting looks promising. However ECPR systems are expensive and resource intensive, making answering this question an imperative.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-70 years old
* Witnessed cardiac arrest
* Bystander CPR
* Refractory cardiac arrest (>20 mins, but <45 mins)
* Initial cardiac rhythm VF, VT or PEA
* Within hours of PACER service operation (e.g. mon-fri 0800-1700)
* Within 25 mins of rapid response ambulance (code 1 lights and sirens)

Exclusion Criteria:

* Initial cardiac rhythm asystole
* ROSC with sustained recovery
* Technically not possible to perform percutaneous cannulation
* Evidence of/suspectedSignificant end stage disease:
* Severe disability impairing activities of daily living
* End-stage organ - cardiac, liver, lung, renal
* Other life-limiting diseases e.g malignancy, terminal illness
* Advance health care directive (not for resuscitation)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in each group that are successfully initiated on ECMO. | 6 months
  Proportion of patients in each group that are successfully initiated on ECMO. This will determine if it is feasible to randomise patients to receive either treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sacha Richardson, MBBS, Principal Investigator — The Alfred

IPD SHARING:
Plan to Share IPD: No